CLINICAL TRIAL: NCT01763983
Title: A Randomized Controlled Trial Testing the Additive Benefits of CBT and Exercise For Psychological Stress and Cognitive Dysfunction in MS
Brief Title: Effects of Cognitive Behavioural Therapy and Exercise on Stress and Cognitive Deficits in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Multiple Sclerosis Society of Canada (Other)
Responsible Party: Principal Investigator, Dr. Neil Rector, Psychologist, Research Scientist and Director of the Mood and Anxiety Treatment and Research Program, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: EG1290
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Multiple Sclerosis; Cognitive Deficits; Stress, Psychological
Keywords: Multiple Sclerosis; Stress, Psychological; Psychological Stress; Emotional Stress; Cognitive Deficits; Cognitive Dysfunction
MeSH Terms: conditions — Multiple Sclerosis; Cognition Disorders; Stress, Psychological; Cognitive Dysfunction | interventions — Cognitive Behavioral Therapy; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aerobic Exercise (Experimental): 12-week structured and monitored aerobic exercise program
  Interventions: Behavioral: Aerobic Exercise
- CBT and Aerobic Exercise (Experimental): Combined 12-week individual Cognitive Behavioural Therapy and Exercise Program
  Interventions: Behavioral: Cognitive Behavioural Therapy; Behavioral: Aerobic Exercise
- Waitlist Condition (No Intervention): 12-week waitlist control condition, after which participants will have the chance to receive CBT group treatment.

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — CBT will be delivered individually, 1 hour per week, for 12 consecutive weeks. CBT for stress in MS is a structured, short-term, present-oriented therapy with an emphasis on problem-solving and the modification of dysfunctional thinking and behaving. Cognitive strategies include the use of dysfunctional thought records for recording and challenging negative automatic thoughts and the use of behavioural strategies to increase involvement and commitment to personal goals.
  Group therapy following a similar protocol (2 hrs/week) will be offered to those in the waitlist condition after completing the study.
  Other Names: CBT
  Arms: CBT and Aerobic Exercise
Behavioral: Aerobic Exercise — Aerobic exercise will occur three times per week at participating gyms. Duration of the exercise periods will be 15-30 minutes for the first 4 weeks (training stage) and 30-45 minutes for the remaining 8 weeks (improvement stage). The exercise regimen will progress from light-moderate exercise (40-60% intensity) to moderate-high exercise (60-80% intensity), following the same course as the increase in duration.
  Arms: Aerobic Exercise; CBT and Aerobic Exercise

SUMMARY:
High levels of psychological stress have been reported by 90% of patients with MS experiencing disease exacerbation, and approximately 39% of those with more stable disease course. These stress levels are comparable to patients with a clinical diagnosis of major depression. Cognitive dysfunction affects approximately 40% of community surveyed MS patients, and stress may exacerbate the cognitive burden. Studies have shown that Cognitive Behavior Therapy (CBT) is effective in treating psychological stress. Studies have also shown that exercise is beneficial to mood and cognitive function. Therefore the proposed study will test the comparative benefits of combining CBT and Exercise as an intervention for stress and cognitive dysfunction in MS subjects. The 2 active treatment conditions will be compared with a waitlist control condition.

There are 4 broad aims to this study: 1) to compare the relative efficacy of CBT, Exercise, and CBT-Exercise for stress in MS, 2) to examine the extent to which neuropsychological features of stress and MS, especially working memory and executive functioning, improve following treatments, 3) to determine the extent to which neuropsychological factors are associated with successful treatment response and improved quality of life, and 4) to determine if combined CBT-Exercise confers greater benefits on measures of stress and neuropsychological functioning compared with Exercise alone.

The study hypotheses are: 1) All active treatment conditions will lead to significantly greater improvement on measures of stress at post-treatment and follow-up compared to waitlist controls, 2) Combined CBT-Exercise will lead to comparatively greater symptom reduction compared to all other conditions at post-treatment and follow-up assessments on measures of stress, 3) All active treatment conditions will lead to significant improvement in neuropsychological functioning (particularly measures of working memory and executive functioning) at post-treatment compared to controls, and 4) Combined CBT-Exercise will lead to greater improvement in neuropsychological functioning compared to all other conditions at post-treatment.

The study design allows for examination of the potential additive benefits of CBT and Exercise to usual therapy for patients, and its feasibility as a viable treatment model for MS outpatient clinics and community-based intervention programs. This study will shed light on the treatment of sub-threshold symptoms that are strikingly common in MS population, but often overlooked in favour of more concrete diagnoses (e.g. major depression disorder). This proposed study will also be the first to determine whether evidence-based non-medical treatments for stress and mood disturbances in MS reduce underlying cognitive substrates associated with the illness and known to be exacerbated by stress.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapse-remitting MS according to the McDonald criteria
* General Health Questionnaire short form (GHQ-12) score of ≥2
* Extended Disability Status Scale (EDSS) score of ≤5
* Physical Activity Readiness Questionnaire (PAR-Q) score of ≤1

Exclusion Criteria:

* Any past history of traumatic brain injury, psychotic mental illness, developmental delay, substance abuse (excluding cannabis) and systemic illness
* Current (last 6 months) participation in an exercise regimen of moderate-strenuous intensity, greater than 2 days a week
* Incapable of providing informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 173 (Actual)
Dates: Start 2013-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in General Health Questionnaire (GHQ-28) at 12 Weeks | Baseline and 12 weeks
  The GHQ-28 is a 28-item self-report used to psychological stress. The GHQ focuses on two main classes of phenomena: 1) inability to carry out one's normal healthy functions; and 2) emergence of new phenomena that are distressing.

SECONDARY OUTCOMES:
Change from Baseline in the Minimal Assessment of Cognitive Function in MS at 12 Weeks | Baseline and 12 Weeks
  The Minimal Assessment of Cognitive Function in MS (MACFIMS)is a 90 minute cognitive battery comprised of seven tests covering five cognitive domains commonly impaired in MS (processing speed/working memory; learning and memory; executive function; visuo-spatial processing; word retrieval).

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada